CLINICAL TRIAL: NCT01793389
Title: Platelet Rich Fibrin in the Treatment of Localized Gingival Recessions: Split-mouth Randomized Clinical Trial
Brief Title: Platelet Rich Fibrin in the Treatment of Localized Gingival Recessions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Gülnihal Eren, Research Asisstant, Dr., Ege University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2010-Dis-002
Record Dates: First submitted 2013-02-12; First posted 2013-02-15 (Estimated); Last update posted 2013-08-15 (Estimated); Status verified 2013-08

CONDITIONS: Gingival Recession
Keywords: gingival recession; fibrin; connective tissue; root coverage; microsurgery; case-control studies
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Subepithelial connective tissue graft (Active Comparator): Soft tissue harvested from palatum of the subjects.
  Interventions: Procedure: Subepithelial connective tissue graft
- Platelet Rich Fibrin (Experimental): Autogenous platelet and leukocyte fibrin material was obtained from blood.
  Interventions: Procedure: Platelet Rich Fibrin

INTERVENTIONS:
Procedure: Subepithelial connective tissue graft
  Arms: Subepithelial connective tissue graft
Procedure: Platelet Rich Fibrin
  Arms: Platelet Rich Fibrin

SUMMARY:
The present study deals with treatment of localized gingival recessions. The hypothesis of this study is that platelet rich fibrin can be used an alternative to subepithelial connective tissue graft in the coverage of denuded roots. If the platelet rich fibrin will prove to be similarly effective as subepithelial connective tissue graft, it will be possible to avoid a donor site and to decrease patient discomfort after operation.

DETAILED DESCRIPTION:
The main objective of this split-mouth, randomized, controlled clinical trial was to compare the clinical efficacy of platelet rich fibrin (PRF) in combination with the coronally advanced flap (CAF) to the use of subepithelial connective tissue graft (SCTG) in combination with CAF in the treatment of localized gingival recessions.

Primary outcome variables were percentage of complete root coverage and change in gingival recession expressed as recession reduction in millimeters at follow-up visits. The secondary outcome variables included keratinized tissue and gingival thickness gain.

Sample size has been estimated in 22 subjects per treatment groups. Random allocation of the treatment sites to test (CAF+ PRF) and control (CAF + SCTG) groups will be performed using a computerized selection of random numbers for allocation of the study groups.

Periodontal parameters including plaque index (25) (PI), gingival index (26) (GI), probing depth (PD), clinical attachment level (CAL), and gingival recession parameters including recession depth (RD), recession width (RW), recession area (RA), keratinized tissue width (KTW), gingival thickness (GT) were assessed by a calibrated examiner. At baseline and 1, 3 and 6 months, RD, RW, RA, KTW were evaluated by means of both clinical and digital assessment. GI and PI were recorded at baseline and 1, 3 and 6 months, however PD, CAL, and GT were evaluated at baseline and 6 months. PD and CAL were recorded by a Williams probe accurate to the nearest 0.5 mm. GT was evaluated at baseline and 6 months using #15 endodontic reamer attached to a rubber stopper inserted perpendicularly into the gingival tissue 2 mm below the gingival margin; thickness was measured to the nearest 0.1 mm using a caliper.

Clinical images obtained at baseline and 1, 3 and 6 months after surgery from each treatment site and digitized in a computer image analysis system. Using a 4-mm length wire was used to check the reproducibility of the pictures. RD was measured from the cement-enamel junction (CEJ) to the gingival margin, RW was measured tangentially at the mid-facial CEJ, RA was calculated as the area within the contour of denuded root. KTW recorded as the distance from the mucogingival junction (MGJ) to the gingival margin. Duplicate measurements were made for RD, RW, RA and KTW. Percent root coverage and complete root coverage was calculated RA according to the following standard formulae.

Follow-up of subjects will be 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Similar bilateral or contralateral Miller Class I or II localized gingival recessions at least ≥ 2 mm located on incisors, canines or premolars on both jaws
* Identifiable CEJ
* Age ≥ 18 years
* Presence of tooth vitality and absence of restorations and superficial caries in the area to be treated
* No periodontal surgical treatment in the previous 24 months on the involved sites
* Gingival thickness at least ≥ 0.8 mm for the recession area
* Sufficient palatal donor tissue for the indicated SCTG.

Exclusion Criteria:

* Smoking
* Patients with a pregnancy or lactation period or self-reported history of antibiotic medication within three months
* Molar, mobile or teeth with crown or filling were also excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2010-01; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Complete root coverage | 1, 3 and 6 months
  Change from baseline in percentage of complete root coverage at 1, 3 and 6 months.
Gingival recession depth | 1, 3 and 6 months
  Change from baseline in gingival recession will be assessed at 1, 3 and 6 months.

SECONDARY OUTCOMES:
Keratinized tissue width | 6 months
  Change from baseline in keratinized tissue at 6 months.
Gingival thickness | 6 months
  Change from baseline in gingival thickness at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Gülnihal Eren, PhD, Principal Investigator — Ege University School of Dentistry; Gül Atilla, Professor, Study Director — Ege University School of Dentistry
Locations (1):
- Ege University School of Dentistry Department of Periodontology, Izmir, Turkey (Türkiye)